CLINICAL TRIAL: NCT00990249
Title: Busulfan Plus Clofarabine Followed by Allogeneic Hematopoietic Stem Cell Transplantation for Patients With Acute Lymphoblastic Leukemia or Lymphoma, or Biphenotypic Leukemia
Brief Title: Busulfan Plus Clofarabine Followed by Allogeneic Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0209; NCI-2012-01270 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-10-02; First posted 2009-10-06 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2017-05

CONDITIONS: Leukemia; Lymphoma; Allogeneic Haematopoietic Stem Cell Transplantation; Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; ALL; Acute lymphoblastic lymphoma; acute biphenotypic leukemia; Allogeneic hematopoietic cell transplantation; HCT; Stem Cell Transplant; Treatment-related mortality; Tyrosine kinase inhibitors; TKI; Busulfan; Busulfex; Myleran; Clofarabine; Clolar; Clofarex; Gleevec; Imatinib Mesylate
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute | interventions — Busulfan; Clofarabine; thymoglobulin; Antilymphocyte Serum; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Busulfan + Clofarabine + Stem Cell Transplant (Experimental): Busulfan test dose 32 mg/m^2 by vein over 45 minutes on Day -8; following doses on Days -6 to -3 derived from pharmacokinetic (PK) testing done up to 11 times over 11 hours after test dose.
  Clofarabine 40 mg/m^2 by vein over 1 hour daily Day -6 through Day -3. Thymoglobulin 0.5 mg/kg on Day -3, 1.5 mg/kg on Day -2 and 2.0 mg/kg on Day -1; only patients with HLA nonidentical or unrelated donors.
  Stem cell infusion on Day 0.
  Interventions: Drug: Busulfan; Drug: Clofarabine; Drug: Thymoglobulin; Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: Busulfan — Test Dose 32 mg/m^2 by vein over 45 minutes on Day -8; following doses on Days -6 to -3 derived from pharmacokinetic (PK) testing done up to 11 times over 11 hours after test dose.
  Other Names: Busulfex; Myleran
Drug: Clofarabine — 40 mg/m^2 by vein over 1 hour daily Day -6 through Day -3
  Other Names: Clolar; Clofarex
Drug: Thymoglobulin — 0.5 mg/kg on Day -3, 1.5 mg/kg on Day -2 and 2.0 mg/kg on Day -1; only patients with HLA nonidentical or unrelated donors
  Other Names: Anti-thymocyte globulin; ATG
Procedure: Stem Cell Transplant — Stem cell infusion on Day 0.
  Other Names: Allogeneic hematopoietic cell transplant; HCT

SUMMARY:
The goal of this clinical research study is to test the safety of giving clofarabine in combination with busulfan, followed by an allogeneic (from a donor) stem cell transplant, in patients with advanced leukemia or lymphoma.

DETAILED DESCRIPTION:
Study Treatment:

Busulfan is designed to bind to DNA (the genetic material of cells), which may cause cancer cells to die. It is commonly used in stem cell transplants.

Clofarabine is designed to interfere with the growth and development of cancer cells.

A stem cell transplant is designed to help your body attack the cancer cells that may remain in your body after chemotherapy.

Central Venous Catheter Placement:

If you are found to be eligible to take part in this study, you will have a central venous catheter (CVC) placed. A CVC is a sterile flexible tube that will be placed into a large vein while you are under local anesthesia. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form for it.

The study drugs and stem cells will be given by vein through your CVC. The CVC will remain in your body for about 3 months.

Study Drug Administration and Stem Cell Transplant:

You will first receive a low-level "test" dose of busulfan by vein, either over 45 or 60 minutes, on Day -8 (8 days before the transplant).

A heparin lock will be placed in your vein to lower the number of needle sticks needed for the blood draws. This will involve placing an intravenous (IV) line in your lower arm that will remain in place from Day -8 through Day -6.

Blood (about 1 teaspoon each time) will be drawn for pharmacokinetic (PK) testing up to 11 times over the 11 hours after the busulfan dose on Day -8. PK testing measures the amount of study drug in the body at different time points. This PK testing will be done to find the dose of busulfan needed for your body size on the other days that you receive busulfan.

Each day from Day -6 through Day -3, you will receive clofarabine by vein over 1 hour and your body-specific dose of busulfan by vein over 3 hours. If for any reason you could not have the PK tests performed, you will receive the standard busulfan dose on these days.

The PK testing will be repeated on Day -6. Blood (about 1 teaspoon each time) will be drawn for PK testing up to 11 times over the 11 hours after the busulfan dose.

If your donor is not related to you or his/her tissue is not HLA-matched (genetically matched), you will receive antithymocyte globulin (ATG) by vein over 4 hours each day on Day -3 through Day -1. ATG is designed to weaken your immune system in order to lower the risk that your body will reject the transplant.

On Day 0, you will receive the donor's bone marrow or blood stem cells by vein. The infusion will last anywhere from about 30 minutes to several hours.

You will also receive tacrolimus and methotrexate to weaken the immune system and lower the risk of graft-versus-host disease (GVHD). GVHD is a reaction of the donor's immune cells against the recipient's body.

* Tacrolimus will be given by vein over 24 hours every day, starting on Day -2 and continuing until you are able to take tacrolimus by mouth. Once you can take tacrolimus by mouth, you will take it every day for about 6 months. If you develop GVHD, the doctor may decide you need to take tacrolimus longer than 6 months.
* Methotrexate will be given by vein over 15 minutes on Days 1, 3, 6, and 11 after the transplant.

Starting 1 week after the transplant, you will receive filgrastim (G-CSF) as an injection under the skin once a day until your blood cell levels return to normal.

Other Possible Treatments:

If you have a history of leukemia or lymphoma in the brain, you will receive spinal taps and chemotherapy several times over the 12 months after the transplant. The chemotherapy drug will be infused over a few minutes, during the spinal tap, directly into the space around the spinal cord. Based on standard care, the doctor will decide how often this occurs and which chemotherapy drug will be used (either methotrexate or cytarabine).

If you have a certain type of leukemia (Philadelphia chromosome positive acute lymphoblastic leukemia [ALL]), you will receive an additional drug to help prevent the cancer from returning. The drug will be imatinib mesylate or another similar type of drug that the doctor decides. It will be given by mouth, every day for up to 1 year after the transplant.

Length of Study Participation:

You will be in the hospital for about 4 weeks after the transplant. You will be taken off study if the disease gets worse. The study drugs will be stopped if intolerable side effects occur.

Follow-Up:

At 1, 3, 6, and 12 months after the transplant, the following tests and procedures will be performed:

* Blood (about 4 tablespoons) will be drawn for routine tests.
* You will have a bone marrow aspiration to check the status of the disease. To collect a bone marrow aspirate, an area of the hip is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle.
* If the disease was not in your bone marrow at the time of diagnosis, you will have a CT and/or positron emission computed tomography (PET) scan to check the status of the disease.

The study staff will stay in contact with your local doctor to find out if the leukemia or lymphoma comes back, as well as to check how you are doing.

This is an investigational study. Busulfan and clofarabine are commercially available and FDA approved for the treatment of cancer. Busulfan is also FDA approved for use with stem cell transplants. The use of these drugs together with a stem cell transplant is investigational.

Up to 150 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with biopsy-proven acute lymphoblastic leukemia, acute lymphoblastic lymphoma, or acute biphenotypic leukemia in remission or relapse.
2. Adequate renal function, as defined by estimated serum creatinine clearance >60 ml/min.
3. Bilirubin equal or less than 1.5 (unless Gilbert's Syndrome), serum glutamate pyruvate transaminase (SGPT) <3 X upper limit of normal and alkaline phosphatase <2 X upper limit of normal.
4. Adequate pulmonary function with forced expiratory volume at one second (FEV1), forced vital capacity (FVC) and diffusion capacity of lung for carbon monoxide (DLCO) at least 45% of expected corrected for hemoglobin. Children unable to perform pulmonary functions must have an oxygen saturation greater than 92% at room air.
5. Adequate cardiac function with left ventricular ejection fraction at least 45% on appropriate medical therapy. No uncontrolled arrhythmias or symptomatic cardiac disease.
6. Zubrod performance status <2 or Lansky/Karnofsky PS equal or greater to 70%.
7. Patients must have a related, genotypically HLA identical donor, or they must have a unrelated donor who is 8/8 HLA match by high resolution typing.
8. Patient or patient's legal representative, parent(s) or guardian should provide written informed consent. Assent of a minor if participant's age is at least seven and less than eighteen years.
9. Negative Beta Human Chorionic Gonadotropin (HCG) test in a woman with child bearing potential defined as not post-menopausal for 12 months and no previous surgical sterilization.

Exclusion Criteria:

1. Patients with unresolved grade >2 non-hematologic toxicity from previous therapy. Patients with grade 2 toxicity will be eligible at the discretion of the PI.
2. Patients with active central nervous system (CNS) disease.
3. Evidence of acute or chronic active hepatitis or cirrhosis.
4. Uncontrolled infection, including HIV, HTLV-1, hepatitis B or hepatitis C viremia.
5. Patients greater than 65 years-old.
6. Prior autologous or allogeneic hematopoietic stem cell transplant.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Partow Kebriaei, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 01, 2009 to July 13, 2015. All recruitment done at The University of Texas MD Anderson Cancer Center.
Groups:
- Busulfan + Clofarabine + Stem Cell Transplant: Busulfan test dose 32 mg/m^2 intravenous (IV) Day -8; following doses Days -6 to -3 derived from pharmacokinetic (PK) testing done up to 11 times over 11 hours after test dose. Clofarabine 40 mg/m^2 IV daily Day -6 through Day -3. Thymoglobulin 0.5 mg/kg Day -3, 1.5 mg/kg Day -2 & 2.0 mg/kg Day -1 for HLA nonidentical or unrelated donors. Stem cell infusion on Day 0.
Period: Overall Study
Arm/Group | Busulfan + Clofarabine + Stem Cell Transplant
Started | 120
Completed | 107
Not Completed | 13
Not completed — Disease Progression | 8
Not completed — Non-Compliance | 1
Not completed — Death | 2
Not completed — Not treated | 2

BASELINE CHARACTERISTICS:
Groups:
- Busulfan + Clofarabine + Stem Cell Transplant: Busulfan test dose 32 mg/m^2 IV Day -8; following doses Days -6 to -3 derived from PK testing. Clofarabine 40 mg/m^2 IV daily Day -6 through Day -3. Thymoglobulin 0.5 mg/kg Day -3, 1.5 mg/kg Day -2 & 2.0 mg/kg Day -1 for HLA nonidentical or unrelated donors. Stem cell infusion on Day 0.
Arm/Group | Busulfan + Clofarabine + Stem Cell Transplant
Number analyzed (Participants) | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 117
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 38 [12 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 86
  Unknown or Not Reported | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 91
  More than one race | 8
  Unknown or Not Reported | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 120

OUTCOME MEASURES:

1. Primary Outcome: Treatment-Related Mortality (TRM) Defined as Non Relapse Mortality (NRM)
Description: NRM was defined as death from any cause other than disease progression or relapse and reported as percentage of participant deaths. Treatment related deaths after transplant are defined either by deaths which could not be attributed to disease relapse or progression or by deaths without previous relapse or progression. For TRM at day 100, Bayesian method of Thall, Simon, and Estey used to perform interim monitoring.
Time Frame: 100 Days
Population: Only 107 participants were evaluated.
Measure: Number; unit: percentage of participants
Arm/Group | Busulfan + Clofarabine + Stem Cell Transplant
Number analyzed (Participants) | 107
percentage of participants | 10

ADVERSE EVENTS:
Time Frame: The specific period was from the start of preparative regiment up to Day 100 for the collection of adverse events.
Arm/Group | Busulfan + Clofarabine + Stem Cell Transplant
Serious Adverse Events (participants affected / at risk) | 3/120
Other Adverse Events (participants affected / at risk) | 118/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Busulfan + Clofarabine + Stem Cell Transplant (N=120)
Diffuse alveolar hemorrhage (DAH) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection/Sepsis (Infections and infestations) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Busulfan + Clofarabine + Stem Cell Transplant (N=120)
Bilirubin (Investigations) | 38 (38)
Transaminitis (Investigations) | 91 (91)
Veno-occlusive disease (VOD) (Vascular disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 56 (56)
Nausea (Gastrointestinal disorders) | 68 (68)
Mucositis (Gastrointestinal disorders) | 105 (105)
Creatinine (Investigations) | 11 (11)
Skin Rash (Skin and subcutaneous tissue disorders) | 22 (22)
Headache (Nervous system disorders) | 6 (6)
Hypertension (HTN) (Vascular disorders) | 16 (16)
Cardiac (Cardiac disorders) | 4 (4)
Fluid Overload (Blood and lymphatic system disorders) | 45 (45)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Shortness of Breath (SOB) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diffuse Alveolar Hemorrahge (DAH) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infection (Infections and infestations) | 92 (248)
Fever (Blood and lymphatic system disorders) | 43 (47)
Neutropenic Fever (Blood and lymphatic system disorders) | 63 (65)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes